CLINICAL TRIAL: NCT01440335
Title: A Study of (R, R') and (S,S': R,R')- Fenoterol: Initial Clinical Evaluation for Pharmacokinetics, Pharmacodynamics, and Safety
Brief Title: Initial Study of Fenoterol as a Treatment for Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 999911153; 11-AG-N153
Record Dates: First submitted 2011-09-23; First posted 2011-09-26 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-01-07

CONDITIONS: Congestive Heart Failure
Keywords: Fenoterol; Pharmacodynamics; Pharmacokinetics; Safety; Beta Adrenergic Agonist
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Drug: Oral R,R'-Fenoterol
Drug: Oral Racemic Fenoterol

SUMMARY:
Background:

- Fenoterol has been used to treat asthma by opening up the airways in the lungs. It also increases the heart rate without significantly increasing blood pressure. This means that it may help improve heart function by boosting the heart's output. Researchers have developed a different form of the drug that may be given to individuals with heart trouble. This new form needs more testing. It is especially important to compare the new form with the original form of the drug used to treat asthma.

Objectives:

- To compare how safe and effective two different forms of Fenoterol are in improving heart function.

Eligibility:

- Healthy people between 21 and 60 years of age who have no history of heart disease.

Design:

* People will be screened with a medical history, physical exam, blood and urine tests, and heart function studies.
* Those in the study will have two 36-hour inpatient study visits. At each visit, they will have a physical exam and blood and urine tests. They will fast overnight and then receive one of the two forms of Fenoterol first thing in the morning. They will not know whether they are getting the original or the modified form of the drug. After receiving the drug, they will provide frequent blood and urine samples for 24 hours. They will have a final exam before being discharged.
* Those who take part in the study will have a followup visit 5 to 7 days after the end of each study visit. They will provide more blood and urine samples and have a physical exam.

DETAILED DESCRIPTION:
Fenoterol is a drug that has been used for the treatment of disease like asthma for many years. It is available in Canada in an inhaled form where it is called Berotec . Fenoterol stimulates receptors in the body called Beta Adrenergic Receptors and is therefore in a family of drugs called Beta Agonists. While one particular form of the drug, called a Racemic mixture has traditionally been used for asthma, multiple forms of the drug have now been produced and it is possible that using one of the newer forms of the drug will have benefits for people with heart failure.

Treatment for heart failure is a complex problem. It is a problem of the heart not pumping enough blood to meet the demands of the body and a number of changes that ultimately prove harmful in an attempt to compensate for this failure. Scientists have observed several effects of Fenoterol that may prove beneficial to people with heart failure. Use of the older Fenoterol (Racemic) mixture indicates that the drug causes the heart to pump more blood out to the rest of the body by increasing a person s heart rate but having little to no effect on their blood pressure. These effects provide a rationale for attempting to develop Fenoterol as a possible treatment for congestive heart failure. It is hoped that this new form of the drug will prove to have even more benefits.

However, the new form of the drug (called the R R form ) has not yet been tested in humans. Animal studies and scientific understanding of these types of mixtures suggest that it will little to no difference between it and the older Racemic form. To test this thinking and determine what doses should be used in future studies, we will conduct a Phase I, escalating dose study in healthy volunteers using the orally administered forms of the older Racemic mixture and newer R R form .

This study will consist of three groups of 6 people taking doses of the drug by mouth and then monitoring their heart rate, blood pressure, blood chemistry, genetic factors, and heart function. The first group will get a 2.5 mg dose of the R R form of the drug on one visit and then a 5 mg dose of the racemic mixture on the other visit. The second group will get a 5mg dose of the R R form on one of their visits and a 10mg dose of the Racemic mixture on the other. Finally, the third group will get a 10mg dose of the R R form on one visit and a 20mg dose of the Racemic mixture on the other. Also, blood will be collected at regular intervals to monitor levels of the drug, its rate of breakdown, changes in blood chemistry, and the testing of various genes. All research will be performed at the National Institute on Aging (NIA) Clinical Research Unit located on the 5th floor of Harbor Hospital in Baltimore, MD.

Testing the safety and breakdown of this drug and comparing it to the older Racemic form will be an important first step in its development as a new drug for heart failure.

The specific aims are:

1. A Phase 1 study in healthy volunteers to establish the body s absorption and breakdown of this new form of Fenoterol (R R form) in comparison with the older, established Racemic mixture.
2. To monitor the effects of the drug on heart rate, blood pressure, and cardiac structure and function after a person takes the drug.

Endpoint: This study will provide a safety assessment and will determine the pharmacokinetics and bioavailability of (R,R )- and racemic Fenoterol in healthy subjects. In addition, information will be gained about the pharmacodynamics of Fenoterol. This will provide information for future studies that will evaluate (R,R )-Fenoterol as a potential treatment for congestive heart failure.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Healthy men and women
2. Age: 21-60
3. Screening laboratory evaluations with no clinically significant abnormal results:

   * Chem-20 panel plus troponin
   * Complete blood count with differential and platelet count
   * Urinalysis with microscopic examination
   * Electrocardiogram
   * Echocardiogram: 2D + Doppler
   * Urine drug screen
   * Urine pregnancy test
4. BMI 24-30
5. Able to provide written informed consent
6. Agree to not participate in other clinical trials during the study period
7. If in child-bearing age and participating in sexual activity that could lead to pregnancy, agree to use a medically accepted method of contraception for a woman for at least 1 month prior to enrollment and continuing 1 month after completion of the fifth study visit, and for a man beginning immediately after the second study visit and continuing for 3 months after completion of the fifth study visit.

EXCLUSION CRITERIA:

1. Resting sitting blood pressure greater than 140/90 mm Hg, resting heart rate greater than 100 bpm
2. Abnormal laboratory examination (ALT and AST greater than 1.5 times the normal range, other labs within 10% of normal range); abnormal troponin screening level will be an exclusion.
3. Clinically significant abnormality on EKG (major Q waves, evidence of heart block, significant conduction disease, QT prolongation)
4. Clinically significant abnormality on Echocardiogram (ejection fraction less than 50 percent, valvular heart disease of moderate severity, pulmonary hypertension with PASP greater than 40mm Hg)
5. Evidence of illicit drug use or alcohol abuse
6. History of Human Immunodeficiency Virus (HIV) infection
7. History of active or chronic Hepatitis B and/or C infection
8. History of malignancy (other than non-invasive skin cancer)
9. History of coronary disease, conduction system disease, pacemaker, atrial fibrillation/flutter, ventricular tachycardia/fibrillation, significant valvular disease, or other cardiovascular disease
10. History of asthma -- reactive airway disease
11. History of seizures or other neurologic diseases
12. History of liver or renal diseases
13. History of gastrointestinal or endocrine disorders (other than mild dyspepsia)
14. Medication use other than occasional use of over-the-counter drugs and/or contraceptives
15. Any medication or herbal drug use within the past 3 days before study participation other than contraceptives
16. Any medical history that, in the opinion of the investigator(s), will make participation of the subject in the study unsafe
17. Participation in another clinical trial involving any pharmacologic agents or blood loss within the past 30 days
18. Donation of blood or blood products within the past 56 days
19. Women who are of childbearing potential and not using acceptable forms of contraception will be excluded.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07-10; Primary Completion 2014-04-15 (Actual); Study Completion 2014-04-15 (Actual)

PRIMARY OUTCOMES:
Safety assessment
Pharmacokinetics
Bioavailability

SECONDARY OUTCOMES:
Pharmacodynamic effects of heart rate
Blood Pressure
Echocardiographic indices of cardiac structure and function
B2-AR lymphocyte binding and function during drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: James B Strait, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Wilson AA, Wang J, Koch P, Walle T. Stereoselective sulphate conjugation of fenoterol by human phenolsulphotransferases. Xenobiotica. 1997 Nov;27(11):1147-54. doi: 10.1080/004982597239903. PMID 9413918
- [Background] Ahmet I, Krawczyk M, Heller P, Moon C, Lakatta EG, Talan MI. Beneficial effects of chronic pharmacological manipulation of beta-adrenoreceptor subtype signaling in rodent dilated ischemic cardiomyopathy. Circulation. 2004 Aug 31;110(9):1083-90. doi: 10.1161/01.CIR.0000139844.15045.F9. Epub 2004 Aug 16. PMID 15313944
- [Background] Anderson G, Wilkins E, Jariwalla AG. Fenoterol in asthma. Br J Dis Chest. 1979 Jan;73(1):81-4. PMID 373786